CLINICAL TRIAL: NCT04619979
Title: Effects of Preoperative Anxiety on Postoperative Outcome and Sleep Quality in Patients Undergoing Laparoscopic Hysterectomy
Brief Title: Preoperative Anxiety on Postoperative Outcome and Sleep Quality in Patients Undergoing Laparoscopic Hysterectomy
Status: Completed | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Other Study IDs: Preoperative anxiety and sleep
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: General Anesthesia; Postoperative Pain; Postoperative Sleep Quality; Preoperative Anxiety
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preoperative anxiety group
  Interventions: Procedure: patients undergoing gynecological surgery under general anesthesia
- Non-preoperative anxiety group
  Interventions: Procedure: patients undergoing gynecological surgery under general anesthesia

INTERVENTIONS:
Procedure: patients undergoing gynecological surgery under general anesthesia — patients undergoing gynecological surgery under general anesthesia

SUMMARY:
Sleep is a naturally occurring state of decreased arousal that is crucial for normal immune and cognitive function. Although surgery and anesthesia techniques have improved in recent years, sleep function and sleep cycles may still be altered perioperatively by surgery and other interventions under general anesthesia.Postoperative sleep fragmentation and poor sleep quality not only lead to hyperalgesia and delayed postoperative recovery, but can increase the risk of potential adverse effects, such as cognitive impairment, chronic pain and emotional disturbances, metabolic disorders, and pro-inflammatory changes. General anesthesia is a medically induced state of hyporesponsiveness that resembles natural sleep. Studies have shown that general anesthesia can lead to circadian rhythm time structure dyssynchrony, resulting in postoperative sleep disturbance, characterized by decreases in rapid eye movement (REM) and slow wave sleep (SWS). Previous studies have also reported that age, preoperative comorbidities, and severity of surgical trauma are independent factors associated with postoperative sleep disturbance. In addition, anxiety is an unpleasant sensation that compromises patients' comfort and well-being. A study by Ruis et al. estimated that 25-80% of patients admitted for surgery experienced preoperative anxiety, including fear of surgery and anesthesia-related fears. Furthermore, preoperative anxiety was recognized as a potential and preventable risk factor for severe postoperative pain and postoperative complications such as increased postoperative morbidity and mortality. Given that several prior studies have reported that preoperative anxiety has an effect on postoperative sleep quality in patients undergoing gynecological surgery, this study aimed to investigate the effect of preoperative anxiety on postoperative outcomes and sleep quality in patients undergoing gynecological surgery. Studying these results could enable us to better manage patients during the perioperative period to promote their postoperative recovery.

ELIGIBILITY:
The inclusion criteria were:

1. age between 18 and 75 years,
2. American Society of Anesthesiologists (ASA) medical status I or II,
3. laparoscopic hysterectomy, elective operation and surgery lasting 1-3 h.

The exclusion criteria included

1. cardiovascular disease,
2. chronic use of analgesics,
3. chronic use of antidepressants,
4. use of sleep-promoting drugs,
5. sleep disorders,
6. sleep apnea syndrome,
7. history of abnormal surgery or recovery from anesthesia,
8. psychosis,
9. patients with impaired verbal communication,
10. unwillingness to provide informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients undergoing gynecological surgery under general anesthesia at Shengjing Hospital of China Medical University.
Sampling Method: Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
postoperative pain | 24 hours after surgery
  evaluate Numerical Rating Scale score (0: no pain to 10: severe pain)
evaluate postoperative sleep quality by using Athens insomnia scale | first night before surgery
  evaluate postoperative sleep by using Athens insomnia scale(<4: no insomnia; 4-6: suspicious insomnia; >6: insomnia)
evaluate postoperative sleep quality by using Athens insomnia scale | first night after surgery
  evaluate postoperative sleep by using Athens insomnia scale (<4: no insomnia; 4-6: suspicious insomnia; >6: insomnia)
evaluate postoperative sleep quality by using Athens insomnia scale | third night after surgery
  evaluate postoperative sleep by using Athens insomnia scale (<4: no insomnia; 4-6: suspicious insomnia; >6: insomnia)
preoperative anxiety score assessed by the Amsterdam preoperative anxiety and information scale (APAIS)". | baseline (before the surgery)
  evaluate the preoperative anxiety score before the surgery, APAIS contains 6 items rated on a five-point Likert scale, which represents two scales: anxiety (items 1, 2, 4, and 5) and need for information (items 3 and 6) Accordingly, the maximal score of the entire APAIS (APAIS-T) is 30 and the one expressing the patient's need for information (APAIS-I) is 10. The maximal score of the two items concerning anxiety about anesthesia (APAIS-A-An) and surgery (APAIS-A-Su) is also 10 each, resulting in a maximal score of 20 for total preoperative anxiety (APAIS-A-T). And APAIS-A-T > 10 was used as a cut-oﬀ to deﬁne patients with high anxiety, the higher the score, the more serious the pre-operative anxiety is

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital, Shenyang, Liaoning, China